CLINICAL TRIAL: NCT00256776
Title: A Randomized Controlled Study of Velcade (Bortezomib) Plus Thalidomide Plus Dexamethasone Compared to Thalidomide Plus Dexamethasone for the Treatment of Myeloma Patients Progressing or Relapsing After Autologous Transplantation
Brief Title: MMVAR - Velcade: Study of Velcade for the Treatment of Myeloma Patients After Autologous Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2005-001628-35; EBMT-CLWP: 42206611
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Results first posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Velcade; Autologous transplantation; Relapse; Disease progress
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib; Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thal + Dex + Velcade (Experimental)
  Interventions: Drug: Velcade (Bortezomib); Drug: Thalidomide; Drug: Dexamethasone
- Thal + Dex (Active Comparator): Standard treatment
  Interventions: Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Velcade (Bortezomib)
  Arms: Thal + Dex + Velcade
Drug: Thalidomide
Drug: Dexamethasone

SUMMARY:
This is an international study in adult patients diagnosed with multiple myeloma who have already received at least one autologous stem cell transplantation and who have responded but later progressed, or relapsed, at least one year after transplantation.

Eligible patients will be randomly assigned to one of two treatments: either Velcade plus Thalidomide plus Dexamethasone or Thalidomide plus Dexamethasone.

Thalidomide and Velcade are two new agents that have recently become available for the treatment of multiple myeloma, especially in relapsed patients. This study therefore aims to test the hypothesis that the combination treatment with Velcade plus Thalidomide plus Dexamethasone will result in a longer time to progression (measure of time after the disease is treated until it starts to get worse) than Thalidomide plus Dexamethasone alone.

DETAILED DESCRIPTION:
Primary Objectives:

* Test the hypothesis that treatment with Velcade plus Thalidomide plus Dexamethasone in combination, will result in a longer time to progression (TTP) than Thalidomide plus Dexamethasone in subjects with relapsed or progressive myeloma after autologous transplantation.

Secondary Objectives:

* Compare the treatment groups for: overall survival; response rate (complete & partial & minimal) using standard criteria and treatment related complications.

Study design and methodology:

This is a prospective, randomized, parallel-group, open-label phase III, on an intention to treat, multicenter study. The main endpoint is time-to-failure (TTP=time to progression). The power is based on an initial assumption of a median TTP of 1.5 years in the experimental (Velcade) group and 1 year in the control group. The design of the study is group sequential. There will be 4 interim analyses and one final analysis. The study is designed to have a priori 90% power to detect the clinically relevant difference at completion of the study at 0.025 level. Patients with multiple myeloma whose disease has either progressed or relapsed at least one year after one or two autologous transplantations will be enrolled. Prior to random assignment, subjects will be stratified on center and number of autologous transplants.Subjects will be randomly assigned to treatment in a 1: 1 allocation within each stratum to Velcade plus Thalidomide plus Dexamethasone (VTD) or Thalidomide plus Dexamethasone. Velcade 1.3 mg/m2 will be given as an i.v. bolus on Days 1, 4, 8 and 11 followed by a 10-day rest period (Days 12 to 21) for 8 cycles (6 months) and then on Days 1, 8, 15, and 22 followed by a 20-day rest period (Days 23 to 42) for 4 cycles (6 months). In both arms, Thalidomide will be given at 200 mg/day per os for one year and Dexamethasone 40 mg/day per os four days every three weeks for one year.Treatment will continue until disease progression, or the occurrence of unacceptable treatment-related toxicity, or up to a total of 12 cycles of Velcade except for those subjects who have a continuing decrease in the levels of paraprotein after 12 cycles. These subjects may continue for as long as treatment is tolerated, and they continue to respond. If a subject has a CR, then treatment should continue at least 2 cycles after the objective response is confirmed. For subjects with a PR or stable disease, treatment may continue after a maximum objective response is confirmed unless the subject experiences unacceptable treatment-related toxicity or the subject has completed 12 cycles of treatment. Disease assessment will occur at the start of each cycle. If a subject discontinues treatment without disease progression, disease assessment will be performed every 3 weeks for 48-weeks from the start of the first dose of study entry drug. Subjects who have not progressed at the end of 48-week follow up period will be assessed every 6 weeks until disease progression is documented

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years-of-age
* Multiple myeloma with evaluable disease
* Relapsing or having a progressive disease
* Karnofsky performance status > 50 %
* Life expectancy of at least 3 months
* Female of child-bearing potential must have a method of birth control and a negative serum or urine beta--human chorionic gonadotropin (β-HCG) pregnancy test at screening and all through the study
* Male must use contraception
* Voluntary written informed consent

Exclusion Criteria:

* Non-secretory multiple myeloma
* Platelet count < 40,000 X 10^9/L
* Absolute neutrophil count <1.0 X 10^9/L
* Creatinine clearance <30 mL/minute
* Peripheral neuropathy >= Grade 2
* Seropositive for HIV, or active hepatitis A, B or C infection
* Pregnant or breastfeeding female
* Patient has hypersensitivity to bortezomib, boron or mannitol
* Other investigational drugs
* Serious medical or psychiatric illness
* Previous or concurrent malignancies at other sites
* Poorly controlled hypertension, uncontrolled or severe cardiovascular disease or uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2005-07; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Garderet, MD, Principal Investigator — Hôpial Saint Antoine, Paris, France - <laurent.garderet@sat.aphp.fr>
Locations (81):
- Austria (4):
  - Karl-Franzens, Graz
  - Universitatsklinik, Innsbruck
  - Medizinische Universitaet Wien, Vienna
  - Wilhelminenspital, Vienna
- Belgium (11):
  - St Joseph, Arlon
  - RHMS, Baudour
  - AZ St Jan, Bruges
  - Bordet, Brussels
  - Erasme CHU, Brussels
  - Saint Luc, Brussels
  - University Hospital, Brussels
  - Saint Joseph, Gilly
  - CH Jolimont, Haine-Saint-Paul
  - Clinique Saint-Pierre, Ottignies
  - UCL Mont-Godinne, Yvoir
- Czechia (2):
  - University Hospital, Brno
  - Faculty Hospital, Olomouc
- France (29):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - Centre Hospitalier d'Antibes, Antibes
  - CHU Jean Minjoz, Besançon
  - Avicenne, Bobigny
  - Polyclinique Bordeaux Nord, Bordeaux
  - Morvan CHU, Brest
  - Hotel Dieu, Clermont-Ferrand
  - ARC CHU Dijon, Dijon
  - Hospitalier de Dunkerque, Dunkirk
  - Hopital Michallon, Grenoble
  - La Roche-sur-Yon
  - Centre Hospitalier du Havre, Le Havre
  - CHRU de Lille, Lille
  - Edouard Herriot, Lyon
  - Pierre Benite, Lyon
  - Metz
  - Centre Hospitalier de Mulhouse, Mulhouse
  - CHU Nancy, Nancy
  - Hotel Dieu, Nantes
  - Archet, Nice
  - Hopital Cochin, Paris
  - Hotel Dieu, Paris
  - Saint Antoine, Paris
  - Hopital Jean Bernard, Poitiers
  - Robert Debre, Reims
  - CHU Hopital Sud, Rennes
  - Henri Becquerel, Rouen
  - CHRU Tours, Tours
- Germany (9):
  - Klinikum Bremen, Bremen
  - University of Cologne, Cologne
  - University Hospital, Dresden
  - University Hospital, Hamburg
  - Medizinische Hochschule, Hanover
  - Uniklinik Leipzig, Leipzig
  - Universitatsklinikum Schleswig-Hostein, Lübeck
  - DKD Wiesbaden, Wiesbaden
  - Medizinische und Poliklinik II, Würzburg
- Hungary (2):
  - St Laszlo Hospital, Budapest
  - University of Debrecen, Debrecen
- Israel (2):
  - Rambam MC, Haifa
  - Sheba MC, Tel Litwinsky
- Italy (9):
  - Ospedale SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ospedale Riuniti, Bergamo
  - AO Spedali Civili di Brescia, Brescia
  - Ospedale Maggiore, Catania
  - Ospedale Maggiore, Milan
  - Federico II, Naples
  - V. Cervello, Palermo
  - Azienda Ospedale BMM, Reggio Calabria
  - A.O.S. Andrea, Rome
- Switzerland (10):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Kantonsspital, Basel
  - IOSI, Ospedale Civico, Bellinzona
  - Inselspital, Bern
  - Hopital Cantonal Universitaire, Geneva
  - CHUV, Lausanne
  - LA Onkologie/Medizin, Thun
  - Stadtdpital Triemli, Zurich
  - UniversitatsSpital, Zurich
- United Kingdom (3):
  - Heartlands Hospital, Birmingham
  - Addenbrookes, Cambridge
  - Great Western Hospital, Swindon

REFERENCES:
- See also: Sponsor's website — http://www.ebmt.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: FPI 08-Jul-2005 LPI 21-Jun-2010
Groups:
- Thal + Dex + Velcade: Velcade (Bortezomib)
  Thalidomide
  Dexamethasone
  Allocated to treatment (n=135) Received allocated treatment (n=135)
- Thal + Dex: Standard treatment
  Thalidomide
  Dexamethasone
  Allocated to treatment (n=134) Received allocated treatment (n=134)
Period: Overall Study
Arm/Group | Thal + Dex + Velcade | Thal + Dex
Started | 135 | 134
Completed | 52 | 54
Not Completed | 83 | 80

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thal + Dex + Velcade | Thal + Dex | Total
Number analyzed (Participants) | 135 | 134 | 269
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 105 | 97 | 202
  >=65 years | 30 | 37 | 67
Age, Continuous [Median (Full Range); unit: years] | 60 [29 to 76] | 62.6 [39 to 75] | 61.2 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 51 | 100
  Male | 86 | 83 | 169
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 5 | 3 | 8
  Belgium | 9 | 14 | 23
  Hungary | 5 | 6 | 11
  Czechia | 5 | 3 | 8
  Italy | 10 | 11 | 21
  United Kingdom | 0 | 1 | 1
  Israel | 1 | 0 | 1
  France | 71 | 68 | 139
  Switzerland | 11 | 8 | 19
  Germany | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression (TTP)
Time Frame: 3 year
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Thal + Dex + Velcade: Velcade (Bortezomib)
  Thalidomide
  Dexamethasone
- Thal + Dex: Standard treatment
  Thalidomide
  Dexamethasone
Arm/Group | Thal + Dex + Velcade | Thal + Dex
Number analyzed (Participants) | 135 | 134
months | 19.5 [16.3 to 22.7] | 13.8 [10.0 to 16.4]

2. Secondary Outcome: Progression Free Survival
Time Frame: 3 year
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Thal + Dex + Velcade: Velcade (Bortezomib)
  Thalidomide
  Dexamethasone
  Median time to progression (primary end point): 19.5 months
- Thal + Dex: Standard treatment
  Thalidomide
  Dexamethasone
  Median time to progression (primary end point): 13.8 months
Arm/Group | Thal + Dex + Velcade | Thal + Dex
Number analyzed (Participants) | 135 | 134
months | 18.3 [15.5 to 20.6] | 13.6 [9.9 to 16.1]

3. Secondary Outcome: Overall Survival (Interval Between Date of Randomization and Death From Any Cause
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Response Rate (Proportion of Subjects Who Achieve Complete, Partial, or Minimal Response)
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Thal + Dex + Velcade | Thal + Dex
Serious Adverse Events (participants affected / at risk) | 58/135 | 45/134
Other Adverse Events (participants affected / at risk) | 0/135 | 0/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thal + Dex + Velcade (N=135) | Thal + Dex (N=134)
Neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Renal Failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Carcinoma (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Vascular Pain (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 7 (7)
Asthenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 16 (21) | 4 (4)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (3)
Various other SAEs (General disorders) | 31 (46) | 30 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No